CLINICAL TRIAL: NCT04982198
Title: Robotic-assisted Versus Conventional Total Knee Arthroplasty: A Multicenter and Randomized Controlled Clinical Trial
Brief Title: Robotic-assisted Versus Conventional Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEA2019-05K
Record Dates: First submitted 2021-07-19; First posted 2021-07-29 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Total Knee Arthoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TKA assisted with ROSA® Knee System (Experimental): TKA assisted with ROSA® Knee System
  Interventions: Procedure: ROSA assisted TKA
- TKA with conventional surgical instrumentation (Active Comparator): TKA with conventional surgical instrumentation
  Interventions: Procedure: ROSA assisted TKA

INTERVENTIONS:
Procedure: ROSA assisted TKA — Robotic assisted total knee arthroplasty

SUMMARY:
This is a multicenter, prospective and randomized controlled pre-market clinical Trial. Study subjects will be randomized into one of two operative groups: 1) TKA assisted with ROSA® Knee System; 2) TKA with conventional surgical instrumentation.

DETAILED DESCRIPTION:
The objective of this clinical trial is to measure the effectiveness and safety of the ROSA® Knee System in assisting surgeons with bone resections and implant positioning optimization through early clinical and radiographic outcomes compared with conventional surgical instrumentation in total knee arthroplasty (TKA).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is age between 18 and 85 years old, inclusive;
2. Patient qualifies for a primary TKA based on the investigator's clinical judgement;
3. Patient is a candidate for commercially available Persona® Knee Joint Prosthese which is compatible with the ROSA® Knee System;
4. Patient is willing and able to provide written Informed Consent.

Exclusion Criteria:

1. Patient planning to receive bilateral TKA surgery within 3 months;
2. Patient who has undergone revision surgery for partial or total knee arthroplasty of the ipsilateral knee；
3. Bone tumor patient who has undergone bilateral TKA;
4. Stable, painless ipsilateral knee arthrodesis within a satisfactory function and position;
5. Patient who has received partial or total knee arthroplasty for the contralateral knee within 6 months prior to scheduled primary TKA;
6. Patient has active, local infection or previous intra-articular infection in the affected joint;
7. Insufficient bone stock on femoral or tibial surfaces;
8. Skeletal immaturity;
9. Osteomalacia or any metabolic disorder which may impair bone formation;
10. Patient has neurologic disorders (e.g. Stroke);
11. Patient hs diseases that could lead to prosthesis instability, failure of prosthesis fixation or postoperative complications (e.g. Arthrodesis, Scoliosis, Lumbar Stenosis)
12. Patient has a hip pathology with significant bone loss (e.g. avascular necrosis of the femoral head with collapse, severe dysplasia of the femoral head or the acetabulum);
13. Patient has hip pathology severely limiting range of motion (e.g. arthrodesis, severe contractures, chronic severe dislocation);
14. Patients with severe knee instability caused by incomplete collateral ligaments, cruciate ligaments, and posterolateral structural injury;
15. Rheumatoid arthritis accompanied by an ulcer of the skin or history of recurrent breakdown of the skin;
16. Patient has severe angular knee deformity of >20° varus or >20° valgus;
17. Patient has a known or suspected sensitivity or allergy to one or more of the implant materials;
18. Patient has other contraindications specified by the implant manufacturer;
19. Patient is pregnant or considered a member of a protected population (e.g. prisoner, mentally incompetent);
20. In the past 1 month participated in or is participating in clinical trials related to other drugs and medical devices;
21. Any other conditions that the investigator considers inappropriate for participation in this trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Mechanical axis alignment | 6 weeks (±2 week) postoperatively
  Deviation from neutral mechanical axis alignment based on full-leg weight-bearing X-ray at 6 weeks (±2 week) postoperatively.

SECONDARY OUTCOMES:
Coronal Lower Limb Alignment | 6 weeks (±2 week) postoperatively
  Coronal Lower Limb Alignment based on full-leg weight-bearing X-ray at 6 weeks (±2 week) postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Yonggang Zhou, Principal Investigator — PLA Hospital
Locations (1):
- PLA Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No